CLINICAL TRIAL: NCT02868190
Title: A Prospective Evaluation of Open-angle Glaucoma Subjects on One Topical Hypotensive Medication (Prostaglandin) Treated With Two Trabecular Micro-bypass Stents (iStent Inject)
Brief Title: Two Second-Generation Trabecular Micro-bypass Stents to Treat Glaucoma Subjects on One Hypotensive Medication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-038
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Two micro-bypass stents (iStent inject) (Other): Standalone implantation of two trabecular micro-bypass stents (iStent inject)
  Interventions: Device: Two trabecular micro-bypass stents (iStent inject)

INTERVENTIONS:
Device: Two trabecular micro-bypass stents (iStent inject) — Standalone implantation of two trabecular micro-bypass stents (iStent inject)

SUMMARY:
This study objective is to evaluate the intraocular pressure (IOP) lowering effect of two trabecular micro-bypass stents (iStent inject) in eyes of subjects with primary open-angle glaucoma on one topical hypotensive medication

DETAILED DESCRIPTION:
The study design is as follows:

Prospective

Subjects with medicated IOP > 18 mmHg and ≤ 30 mmHg

Subjects on one topical ocular hypotensive medication prior to stent implantation

Implantation of two iStent devices (if IOP is < 6 mmHg, at any point during the postoperative follow-up, medication will not be prescribed or will be discontinued)

IOP will be measured by two (2) observers to minimize bias; observer 1 will look through the slit lamp and turn the dial with readings being masked, and observer 2 will document the IOP

Diurnal IOP measurements

Follow-up through 60 months postoperative (but could be up to 61 months if subject needs to undergo terminal washout)

Descriptive statistics will be tabulated

Medical therapy considered necessary for the subject's welfare can be implemented at any time during the study at the investigator's discretion

ELIGIBILITY:
INCLUSION CRITERIA:

Screening Exam Inclusion Criteria:

* Phakic patients or pseudophakic patients with posterior chamber intraocular lenses (PC-IOLs).
* Primary open-angle glaucoma (including pigmentary or pseudoexfoliative).
* Cup-to-disc ratio ≤ 0.9.
* Visual field defects, or nerve abnormality characteristic of glaucoma.
* One topical hypotensive medication at time of screening exam.
* Intraocular pressure (IOP) > 18 mmHg and ≤ 30 mmHg (medicated) at screening exam.
* Study eye BCVA 20/100 or better.
* Normal angle anatomy as determined by gonioscopy.
* Absence of peripheral anterior synechia (PAS), rubeosis or other angle abnormalities that could impair proper placement of stent.

Baseline Exam Inclusion Criteria:

* Subject has completed appropriate medication washout.
* Mean IOP > 22 mmHg and ≤ 38 mmHg after anti-glaucoma medication washout period.

EXCLUSION CRITERIA:

Screening Exam Exclusion Criteria:

* Aphakic patients or pseudophakic patients with anterior chamber IOLs (AC-IOLs).
* Prior stent implantations (study eye).
* Traumatic, uveitic, neovascular, or angle-closure glaucoma; or glaucoma associated with vascular disorders.
* Functionally significant visual field loss, including severe nerve fiber bundle defects such as Bjerrum scotoma.
* Prior incisional glaucoma surgery.
* Prior SLT within 90 days prior to screening.
* Prior ALT.
* Iridectomy or laser iridotomy.
* Ineligibility for ocular hypotensive medication washout period as determined by the investigator such as: visual field status would be placed at risk by washout period, or unmedicated IOP after washout period would be expected to exceed upper limit of ≥ 38 mmHg.
* Any active corneal inflammation or edema (e.g., keratitis, keratoconjunctivitis, keratouveitis).
* Clinically significant corneal dystrophy (e.g., bullous keratopathy, Fuch's dystrophy); any guttata.
* Corneal surgery (prior or anticipated) of any type (including LASIK, LASEK, PRK, etc.) that may interfere with IOP measurement reliability.
* Corneal opacities or disorders that would inhibit visualization of the nasal angle.
* Congenital or traumatic cataract.
* Retinal or optic nerve disorders, either degenerative or evolutive, that are not associated with the existing glaucoma condition.
* Elevated episcleral venous pressure such as associated with: active thyroid orbitopathy, cavernous sinus fistula, Sturge-Weber syndrome, orbital tumors, orbital congestive disease.
* Clinically significant sequelae from trauma (e.g., chemical burns, blunt trauma, etc.).
* Chronic ocular inflammatory disease or presence of active ocular inflammation (e.g., uveitis, iritis, iridocyclitis, retinitis).
* Pregnant or nursing women.

Baseline Exam Exclusion Criteria:

* Subject did not complete medication washout.
* Mean IOP < 22 mmHg or > 38 mmHg after anti-glaucoma medication washout.
* Subject did not have a 3mmHg IOP increase over screening mean diurnal IOP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Mean intraocular pressure reduction of 20% or more vs baseline | 12 months post-op

SECONDARY OUTCOMES:
Proportion of subjects with intraocular pressure less than or equal to 18 mm Hg | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lilit Voskanyan, MD, PhD, Principal Investigator — S.V. Malayan Eye Center
Locations (1):
- S.V. Malayan's Ophtalmology Centre, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindstrom R, Lewis R, Hornbeak DM, Voskanyan L, Giamporcaro JE, Hovanesian J, Sarkisian S. Outcomes Following Implantation of Two Second-Generation Trabecular Micro-Bypass Stents in Patients with Open-Angle Glaucoma on One Medication: 18-Month Follow-Up. Adv Ther. 2016 Nov;33(11):2082-2090. doi: 10.1007/s12325-016-0420-8. Epub 2016 Oct 13. PMID 27739003
- [Derived] Lindstrom R, Sarkisian SR, Lewis R, Hovanesian J, Voskanyan L. Four-Year Outcomes of Two Second-Generation Trabecular Micro-Bypass Stents in Patients with Open-Angle Glaucoma on One Medication. Clin Ophthalmol. 2020 Jan 13;14:71-80. doi: 10.2147/OPTH.S235293. eCollection 2020. PMID 32021070